CLINICAL TRIAL: NCT02644330
Title: A Randomized Controlled Trial of Minimally Invasive Transthoracic Device Closure in the Treatment of Patients With Perimembranous Ventricular Septal Defect
Brief Title: Minimally Invasive Transthoracic Device Closure in Perimembranous Ventricular Septal Defect
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Associate chief physician in pediatric cardiac surgery, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-ZH39
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Perimembranous Ventricular Septal Defect
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgical group (Active Comparator): The patients in Group A (surgical group) underwent surgical repair with cardiopulmonary bypass
  Interventions: Procedure: surgical repair
- closure group (Experimental): The patients in Group B (closure group) underwent minimally invasive transthoracic device closure.
  Interventions: Procedure: transthoracic device closure

INTERVENTIONS:
Procedure: transthoracic device closure — minimally invasive transthoracic device closure
  Arms: closure group
Procedure: surgical repair — surgical repair with cardiopulmonary bypass
  Arms: surgical group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of minimally invasive transthoracic device closure of ventricular septal defect. This is a multi-center randomized controlled trial. Because of the characteristics of this surgical clinical trials, surgeons, ultrasonic department doctors, anesthesiologists, operating room nurses and intensive care unit nurses are all need to be informed. Therefore the results of this trial need to be system evaluated through objective methods to reduce bias.

DETAILED DESCRIPTION:
Several examinations need to be done in all the patients, including X-ray, electrocardiogram, echocardiogram, blood routine examination, liver and kidney function, electrolytes, coagulation function and infectious index checks. And they will be divided into two groups after they have obtained informed consent: surgical group (50 cases); closure group (50 cases). If the closure failed, the patients in closure group will be converted to surgical repair with cardiopulmonary bypass .

Recheck X-ray, electrocardiogram, echocardiogram, blood routine examination, liver and kidney function and electrolytes need to be done in all the patients two days after operation. The patients were followed up by X-ray, electrocardiogram, echocardiogram at the first month, third month, sixth month and the first year.

ELIGIBILITY:
Inclusion Criteria:

* Age≥3 months
* Patients with isolated perimembranous ventricular septal defect with hemodynamic abnormalities. Diameter of the defect is greater than 3mm, and less than 10mm

Exclusion Criteria:

* Para adverse ventricular septal defect
* Muscular ventricular septal defect, subpulmonic ventricular septal defect and septal leaflet posterior atrioventricular canal ventricular septal defect
* Patients with severe pulmonary hypertension in right-to-left shunt
* Patients with obvious aortic valve prolapse, with moderate or severe aortic regurgitation
* Infective endocarditis, and heart cavity neoplasm
* Patients with other cardiovascular malformations, which require surgery with cardiopulmonary bypass to correct at the same period

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
the success rate of the operation | index procedure (day 0)
  The definition of a successful operation: shunt disappeared

SECONDARY OUTCOMES:
adverse events | 12 months
  death, cardiac perforation, cardiac tamponade, emerging tricuspid regurgitation, emerging aortic regurgitation, arrhythmias (third-degree atrioventricular block, complete bundle branch block), postoperative residual shunt (refers to the residual shunt, which diameter greater than 2mm or flow rate greater than 3m/s), infective endocarditis, postoperative murmur
thoracic fluid volume | index procedure (day 0)
blood transfusion | index procedure (day 0)
operating time | index procedure (day 0)
  time cost from cut the skin to complete closure of the sternum
postoperative ventilator support time | index procedure (day 0)
postoperative hospital stay | 7 days after operation or before discharge
costs | 7 days after operation or before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, Dr, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (3):
- China (3):
  - Henan Province People's Hospital, Zhengzhou, Henan
  - XiangYa Hospital CentralSouth University, Changsha, Hunan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan